CLINICAL TRIAL: NCT02227628
Title: Absorption and Antioxidant Effects of Polyphenolics From Acai
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TexasAMU-IRB2010-0797F; IRB2010-0797F (Other: Texas AMU)
Record Dates: First submitted 2014-06-04; First posted 2014-08-28 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Cardiovascular Disease; Metabolic Syndrome; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Syndrome; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugary Beverage (Placebo Comparator): Sugary Beverage
  Interventions: Dietary Supplement: Sugary Beverage
- Acai beverage (Experimental): Acai Polyphenolics
  Interventions: Dietary Supplement: Acai polyphenolics

INTERVENTIONS:
Dietary Supplement: Acai polyphenolics — Acai beverage was obtained from the Sambazon (San Clemente, CA).
  Arms: Acai beverage
Dietary Supplement: Sugary Beverage — An equal amount of placebo juice comprised of artificially colored water containing sugar (5%), citric acid (0.01% to adjust the pH 3.8), and artificial colors (FD&C Red 40 and Blue 1, Tetra Pak, Denten, TX) that was identical to the acai beverage.
  Arms: Sugary Beverage

SUMMARY:
A human clinical consumption trial will be performed in volunteers with increased risk factors for cardiovascular disease (Metabolic Syndrome), which includes obesity and diabetes and related conditions over a period of 12 weeks with blood draws at baseline (0 weeks), 4, 8, and 12 weeks and a 24 hr urine collection on each blood draw day.

DETAILED DESCRIPTION:
1. Experimental Design: Approximately 50 male and female participants between the ages of 18 and 65 years, who were at high risk for cardiovascular disease but have not had a hospitalization due to cardiovascular disease, were recruited to participate for 12 weeks in this study. All familiarization and testing were conducted at the Exercise & Sport Nutrition Laboratory (ESNL) in the Department of Health and Kinesiology at Texas A&M University. Assays were conducted at the Institute of Obesity and Cancer research Laboratory at Texas A&M University.
2. Screening and familiarization Session:

   Participants expressing interest in the study were interviewed by phone to determine whether they were qualified to participate. The participants who were believed to meet the eligibility criteria were invited to attend an entry/familiarization session. During this session, participants completed medical and personal histories, and signed consent statements in compliance with the Human Participants Guidelines of Texas A&M University and the American College of Sports Medicine. Participants then underwent a general physical examination to verify that they met the eligibility criteria. Participants who satisfied the criteria were familiarized to the study protocol and received a verbal and written explanation of the study protocol and design. Following baseline measurements, participants were matched based on gender, age, and BMI and were randomly assigned in a double-blind manner into control (n=25) or acai supplementation groups (n=25). Participants were given an appointment time to perform baseline assessments and three other sessions.
3. Baseline assessments and dietary intervention:

   Prior to baseline testing, participants were recommended not to take any herbal supplements or anti-oxidant juices such as orange, pomegranate, or acai juice. Vitamin pills, supplemented sports/energy drinks and large amounts of berries were also to be avoided. In addition, spinach, tomatoes, bell peppers, onions, garlic, carrots, chocolate, yellow/orange fruits/vegetables and dark green fruits/vegetables were to be reduced to no more than one serving for 48 hours. Participants were instructed to refrain from exercise for 48 hours prior to baseline testing. During the baseline testing, participants recorded all food intake on dietary record forms for four days. Participants donated 20ml of fasting blood using venipuncture techniques of an antecubital vein in the forearm. Participants were then asked to drink one 10 oz serving of the test beverage. A second blood draw was taken two hours after ingestion. All urine output for the 24 hours leading up to the baseline testing was collected.
4. Supplementation:

   Participants were recommended to consume two servings of the test beverage as part of their current, non-modified diet. Each serving was supplied in a 10 oz bottle, and was to be consumed both in the morning and in the evening of each day throughout the duration of the study (12 weeks). Participants in the control group consumed an equal amount of placebo juice comprised of artificially colored water containing sugar, citric acid, and a flavor that was identical to the acai beverage, but had no phytochemical-based constituents throughout the same time period. Participants were individually instructed on how to adjust their daily caloric intake to account for the calories of the beverage. All participants picked up weekly supplies of either the acai beverage or placebo at the Exercise & Sport Nutrition Laboratory.
5. Follow-up testing:

   Participants reported back to the lab for follow-up testing at 4, 8, and 12 weeks after the baseline testing. During each of those testing sessions, the participants completed the same full battery of tests that were completed during the initial baseline testing. Participants were asked to maintain a similar diet three days prior to each testing session in order to monitor the influence of the test beverage. Participants were given a list of preferred food groups for these three days and asked to stick to them as closely as possible.
6. Body composition:

   During each baseline measurement and follow-up testing session, height was measured using standard anthropometry. Total body weight was measured using a Healthometer (Bridgeview, IL) self-calibrating digital scale with a precision of +/-0.02 kg. Body composition (excluding the cranium) was determined using a Dual-energy X-ray absorptiometry (DEXA, Hologic Inc, Waltham, MA, USA).
7. Blood and urine collection: During each of the testing sessions, participants donated approximately 2 teaspoons of fasting venous blood (10 milliliters). Blood samples were obtained using standard phlebotomy procedures using standard sterile venipuncture of an antecubital vein by ESNL laboratory technicians or graduate research assistance trained in phlebotomy in compliance with guidelines established by the Texas Department of Health and Human Services.

ELIGIBILITY:
Inclusion Criteria:

* Elevated waist circumference: ≥102cm in men and ≥ 88 cm in women
* Elevated triglycerides:≥ 150 mg/dL
* Reduced HDL-C:<40 mg/dL in men and <50 mg/dL in women
* Elevated blood pressure:≥ 130 mmHg systolic blood pressure or ≥ 85 mmHg diastolic blood pressure
* Elevated fasting glucose:≥ 100 mg/dL

Exclusion Criteria:

* History of any relevant acute cardiac event (myocardial infarction, episode of heart failure)
* Recent (within 3 months) or recurrent hospitalizations
* Drug treatment for type II diabetes
* aspartate aminotransferase or alanine aminotransferase ≥ 2 times the upper limit of normal
* Abuse of alcohol or substance, smoking, history of seizures, or other relevant ongoing or recurrent illness, liver or renal dysfunction, pregnancy (positive urine pregnancy test) or lactation, known allergy against any of the juices, known infection with hepatitis B, C, or HIV, intake of vasoactive drugs
* Individuals participating in regular aerobic exercise training program (>30 minutes, ≥ 3 times/wk)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in the levels of Inflammatory biomarkers in plasma or urine | baseline, 24 hours
  During each of the testing sessions, participants donated approximately 2 teaspoons of fasting venous blood (10 milliliters). All urine output for the 24 hours leading up to the baseline testing was collected. Inflammatory biomarkers in the plasma (hs-C-reactive protein(mg/L), interleukin-6(pg/ml), interleukin-1beta(pg/ml), Interferon-gamma(pg/ml), and Tumor necrosis factor-alpha(pg/ml)) and in the urine (8-isoprostane(ng/mmol creatinine) were measured by enzyme immunoassay using Cayman chemical kits (Ann Arbor, MI).

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Talcott, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Exercise & Sport Nutrition Laboratory (ESNL) in the Department of Health and Kinesiology at Texas A&M University, College Station, Texas, United States